CLINICAL TRIAL: NCT02787798
Title: Evaluation of the Effect of Double Inhibition of Angiotensin II AT1 Receptor and Neprilysin Activity on Sympathic Nervous System Activity in Patient With Heart Failure
Brief Title: Evaluation of the Entresto Effect on Sympathic Nervous System in Patient With Heart Failure
Acronym: B2AN-SNS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Today Entresto treatment has marketing authorization and is available for all patients, that is the reason why study was halted prematurely.
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC31/15/7746
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
Keywords: Nervous System; Cardiac disease
MeSH Terms: conditions — Heart Failure; Neurologic Manifestations; Heart Diseases | interventions — Valsartan; sacubitril; sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Entresto (Experimental): * Stop of all angiotensin-converting-enzyme inhibitor or antagonist of angiotensin II receptor during 2 days.
  * valsartan/sacubitril 100 mg tablets (51 and 49 mg) during 2 to 4 weeks twice a day.
  * valsartan/sacubitril 200 mg tablets (103 and 97 mg) during 2 to 4 weeks twice a day.
  * Microneurography recording of sympathetic activity in muscle destiny (MSNA)
  Interventions: Drug: valsartan/sacubitril 100 mg; Drug: valsartan/sacubitril 200 mg; Procedure: Microneurography
- Control (Placebo Comparator): * Hearth failure treatment as usual (angiotensin-converting-enzyme inhibitor or antagonist of angiotensin II receptor)
  * Microneurography recording of sympathetic activity in muscle destiny (MSNA) will be done
  Interventions: Procedure: Microneurography

INTERVENTIONS:
Drug: valsartan/sacubitril 100 mg — Treatment with 100 mg tablets during 2 to 4 weeks
  Other Names: Entresto 100 mg
  Arms: Entresto
Drug: valsartan/sacubitril 200 mg — Treatment with 200 mg tablets during 2 to 4 weeks
  Other Names: Entresto 200 mg
  Arms: Entresto
Procedure: Microneurography — Microneurography recording of sympathetic nervous system activity in muscle destiny
  Other Names: MSNA

SUMMARY:
The hyperactivation of the sympathetic nervous system is a feature of the heart failure and the determinants of disease progression and risk of sudden cardiac death. This research project aims to study, in the drug use conditions provided in the summary of product characteristics based on European marketing authorization (indications and dosage), the effect of the Entresto® on the activity of sympathic nervous system using the reference method, the microneurographic recording of sympathetic activity in muscle destiny (MSNA). This study will try to determine if the double inhibition of AT1 receptor and neprilysin activity result in lower sympathic nervous system burst rate versus single AT1 receptor inhibition using angiotensin-converting-enzyme inhibitor or AT1 receptor of angiotensin II inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Men or women with heart failure with symptomatic left ventricular systolic dysfunction (left ventricular ejection fraction ≤ 40 %) with :

  * Functional class New York Heart Association II and at least 2 hospitalizations for cardiac decompensation in the year with N terminal pro brain-type natriuretic peptide ≥300 pg/ml (or brain-type natriuretic peptide ≥100 pg/ml) or usage of intravenous diuretics,
  * Functional class New York Heart Association III-IV,
  * Insufficiently controlled by alternative drug-free therapies (surgery, cardiac resynchronization ...) or well managed drug therapies: angiotensin-converting-enzyme inhibitor, AT1 receptor of angiotensin II inhibitor diuretics or beta blockers.
  * Treated by maximum dosage of AT1 receptor of angiotensin II inhibitor or angiotensin-converting-enzyme inhibitor for New York Heart Association II patient or 50% of the recommended dose for New York Heart Association III-IV patients or New York Heart Association II patients with clinical manifestation restricting the use of maximum dosage, like orthostatic hypotension.
* Patient member of his home social security scheme

Exclusion Criteria:

* Patient who are receiving direct renin inhibitor like aliskiren
* Patient who are receiving phosphodiesterase V inhibitors
* Patient who are receiving a potassium-sparing drug
* Patient with medical history of angioedema with previous treatment by angiotensin-converting-enzyme inhibitor or AT1 receptor of angiotensin II inhibitor
* Hypersensitivity to any component of Entresto®
* Adult protected by the law
* Severe renal impairment (DFGe <30 ml/min/1,73 m2)
* Severe hepatic impairment, cirrhosis or cholestasis (Child-Pugh C class)
* Patient with are receiving anticoagulant therapies or suffering from known hemostatic trouble
* Patient participating in another biomedical research or with an active exclusion period
* Pregnancy
* Breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of sympathetic nervous system activity as assessed by microneurography recording recording of sympathetic activity in muscle destiny | Up to 8 weeks
  Evaluation of sympathetic nervous system activity in burst/minute

SECONDARY OUTCOMES:
Evaluation of severity of heart failure | Day 0
  assessed by New York Heart Association stage
Evaluation of severity of heart failure | Day 2
  assessed by New York Heart Association stage
Evaluation of severity of heart failure | Up to 4 weeks
  assessed by New York Heart Association stage
Evaluation of severity of heart failure | Up to 8 weeks
  assessed by New York Heart Association stage
Comparison of treatment effect on pro-brain natriuretic peptide serum levels at baseline and at the end of treatment period | Day 0 and up to 8 weeks
  pro-brain natriuretic peptide serum levels

CONTACTS AND LOCATIONS:
Overall Officials: Michel Galinier, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided